CLINICAL TRIAL: NCT06714643
Title: Antidepressant and Related Neurophysiological Effects of Non-invasive Brain Stimulation in Subjects with Major Depressive Disorder
Brief Title: Non-invasive Brain Stimulation in Subjects with Major Depressive Disorder
Acronym: NIBS_tDCS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Carmen Concerto (Other)
Responsible Party: Sponsor-Investigator, Carmen Concerto, PhD, MD, University of Catania
Organization: University of Catania (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 130/2022/PO
Record Dates: First submitted 2024-09-16; First posted 2024-12-03 (Actual); Last update posted 2024-12-03 (Actual); Status verified 2024-11

CONDITIONS: Major Depressive Disorder (MDD)
Keywords: tDCS; MD; Biomarkers
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- active (Experimental)
  Interventions: Device: Active tDCS
- sham (Sham Comparator)
  Interventions: Device: Sham treatment

INTERVENTIONS:
Device: Active tDCS — The active tDCS protocol consist of 15 excitatory tDCS sessions distributed over 3 weeks (5 sessions per week, from Monday to Friday), at the same time each day, administered by the same operators and under identical experimental conditions. Each session last 30 minutes, with the Anode electrode placed on the left dorsal lateral prefrontal cortex (DLPFC) and the Cathode electrode on the right DLPFC at an intensity of 2 mA. The electrodes are positioned according to the 10-20 electroencephalography system (Anode on F3 and Cathode on F4).
  Arms: active
Device: Sham treatment — The sham-tDCS intervention consist of a placebo 15 tDCS sessions distributed over 3 weeks (5 sessions per week, from Monday to Friday), at the same time each day, administered by the same operators and under identical experimental conditions. Each session last 30 minutes, with the Anode electrode placed on the left dorsal lateral prefrontal cortex (DLPFC) and the Cathode electrode on the right DLPFC. During the sessions only a 15-second initiation current is applied, providing the patient with the sensation of receiving an electric current on the scalp. Participants will also experience sounds and stimuli similar to those produced by active tDCS.
  Arms: sham

SUMMARY:
Introduction The study involves the recruitment of outpatients suffering from Major Depressive Disorder (MDD), diagnosed according to the criteria of the Diagnostic and Statistical Manual of Mental Disorders (DSM-5). Patients are on selective serotonin reuptake inhibitors (SSRIs) for at least 4 weeks and present residual depressive symptoms, defined by a score greater than 7 on the Hamilton Depression Rating Scale (HDRS-17).

Study Objectives

Primary Objective To investigate the effects of transcranial direct current stimulation (tDCS) on depressive symptoms in patients with depression, randomized into a "test" group and a "sham" group.

Secondary Objectives

To investigate the effects of tDCS on cognitive function in patients with depression, randomized into a "test" group and a "sham" group.

To evaluate changes in blood biomarkers, neurophysiological, and neurosonological variables after tDCS treatment in the same group of patients.

ELIGIBILITY:
Inclusion criteria:

* Patients with Major Depressive Disorder (MDD), as defined by the DSM-5-TR criteria;
* Presence of residual symptoms, defined by a Hamilton Depression Rating Scale score over 7;
* Age over 18 years.

Exclusion criteria:

* MMSE under 18 and/or CDR over 2;
* Other neurological diseases (stroke, multiple sclerosis, major head trauma, epilepsy) or psychiatric disorders other than those included (schizophrenia, bipolar disorder, etc.);
* Patients with severe clinical conditions, acute or uncontrolled chronic medical diseases;
* Endocrine diseases, vitamin deficiencies, or exposure to drugs associated with cognitive impairment and/or mood deflection;
* Alcohol abuse or recreational drug use;
* Contraindications to MRI and TMS (carriers of implanted devices, patients who have undergone craniotomy, presence of metal fragments or prostheses, history of epilepsy);
* Pregnant or breastfeeding women.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Estimated)
Dates: Start 2025-01-02 (Estimated); Primary Completion 2026-01-02 (Estimated); Study Completion 2026-01-02 (Estimated)

PRIMARY OUTCOMES:
Hamilton Depression Rating Scale - 17 (HDRS-17) | From enrollment to the end of treatment at 6 months
  To investigate the effects of transcranial direct current stimulation (tDCS) treatment by administering Hamilton Depression Rating Scale - 17 (HDRS-17) on depressive symptoms in patients with depression, randomized into a "test" group and a "sham" group. Higher scores indicate greater severity of depressive symptoms, and thus a worse outcome.
  The minimum and maximum scores and their meaning are as follows: 0-7: No clinically significant depression; 8-13: mild depression; 14-18: moderate depression; 19-22: severe depression; 23-52: very severe depression.

SECONDARY OUTCOMES:
Montreal Cognitive Assessment (MOCA) | From enrollment to the end of treatment at 6 months
  To investigate the effects of tDCS treatment on cognitive function in patients with depression, randomized into a "test" group and a "sham" group.
  Lower scores suggest greater cognitive impairment, while higher scores indicate better cognitive performance. Below are the minimum and maximum scores and their meaning: 30-26: normal cognitive function; 25-18: mild cognitive impairment; 17-10: moderate cognitive impairment; 9-0: severe cognitive impairment.
Frontal Assessment Battery (FAB) | From enrollment to the end of treatment at 6 months
  To investigate the effects of tDCS treatment on cognitive function in patients with depression, randomized into a "test" group and a "sham" group. Specifically, FAB is a tool used to evaluate frontal lobe functions, such as executive functioning. Lower scores suggest greater impairment of frontal lobe functions, while higher scores indicate better functioning. Below are the minimum and maximum scores and their meaning: 18-15: normal frontal lobe functioning; 14-12: mild impairment; 11-9: moderate impairment; 9-0: severe impairment.
Apathy Evaluation Scale (AS) | From enrollment to the end of treatment at 6 months
  To investigate the effects of tDCS treatment on cognitive function in patients with depression, randomized into a "test" group and a "sham" group. AS is a tool used to assess the presence of apathy in patients. Higher scores suggest greater severity of apathy, while lower scores indicate better motivation and engagement. Below are the minimum and maximum scores and their meaning: 18-27: no clinically significant apathy; 28-41: mild apathy; 42-55: moderate apathy; 56-72: severe apathy.
Stroop Color Test | From enrollment to the end of treatment at 6 months
  To investigate the effects of tDCS treatment on cognitive function in patients with depression, randomized into a "test" group and a "sham" group. Stroop Color Test is a neuropsychological tool used to assess cognitive flexibility, selective attention and processing speed. Performance is assessed by comparing raw scores to normative data adjusted for age, education and cultural background. Minimum score (0) indicates no ability to perform the task; on the other hand, there is no universal maximum score. Tipically, performance is categorized into a normal range when it is consistent with age-matched norms; mild impairment when the performance is slightly below expectations for age or education; moderate to severe impairment when patient shows significant difficulty with cognitive control or selective attention.
To evaluate changes in blood biomarkers after tDCS treatment | From enrollment to the end of treatment at 6 months
  A blood sample is collected at enrollment and after tDCS/sham treatment to evaluate biomarkers, including BDNF, NGF, VEGF, IGF1, Ang, Nrg1, IL-6, and TNFα.
  Concentrations will be reported in pg/mL or ng/mL, as appropriate for each biomarker.
To evaluate changes in cerebral hemodynamics after tDCS treatment | From enrollment to the end of treatment at 6 months
  A transcranial Doppler (TCD) exam is conducted to assess cerebral hemodynamics. Parameters including VPS (cm/s), EDV (cm/s), MBFV (cm/s), PI (unitless), and RI (unitless) are recorded bilaterally from the middle cerebral arteries and the basilar artery, both at rest and after breath-holding tests. Measurements will be reported in their respective units (e.g., cm/s for velocities, unitless for indices).
To evaluate changes in Cortical Excitability Using TMS | From enrollment to the end of treatment at 6 months
  Cortical excitability is evaluated using transcranial magnetic stimulation (TMS) with single- and double-pulse protocols. Parameters include:
  Resting motor threshold (rMT, % of maximum stimulator output); Cortical silent period (cSP, milliseconds); Motor evoked potential (MEP, µV); Paired-pulse stimulation (BiSTIM) is used to study inhibitory and excitatory circuits, including intracortical inhibition (ICI) and intracortical facilitation (ICF).
  Results are reported in their respective units (e.g., % stimulator output for rMT, ms for cSP, µV for MEP).

CONTACTS AND LOCATIONS:
Overall Officials: Maria Salvina Signorelli, MD PhD, Principal Investigator — University of Catania

IPD SHARING:
Plan to Share IPD: Undecided